CLINICAL TRIAL: NCT05545956
Title: Analysis of Red Blood Cell Integrity and Efficiency of Recovery Using a Novel Surgical Sponge-Blood Recovery Device (ProCell): Delayed Impact
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due staffing issues
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: ProCell Surgical Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY20220888_2
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Blood Recovery
Keywords: Open Heart Surgery; Heart Transplant; Lung Transplant; ProCell

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hand Wrung (Active Comparator): Hand wrung refers to manually wringing surgical sponges by hand.
  Interventions: Procedure: Hand Wrung
- ProCell Wrung (Experimental): ProCell wrung refers to automated wringing surgical sponges by an FDA approved suction device (ProCell).
  Interventions: Device: ProCell Wrung

INTERVENTIONS:
Procedure: Hand Wrung — Hand wrung refers to manually wringing surgical sponges by hand.
  Arms: Hand Wrung
Device: ProCell Wrung — ProCell wrung refers to automated wringing surgical sponges by an FDA approved suction device (ProCell).
  Arms: ProCell Wrung

SUMMARY:
The purpose of this research study is to compare two methods of recovering blood from surgical sponges used during heart and lung surgeries. The two methods are: 1) manually wringing sponges by hand, and 2) automated wringing sponges by an FDA approved suction device. Both methods are already in use in heart and lung surgeries at University Hospitals at the discretion of the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing heart or lung transplant, redo sternotomy, aortic surgery, and/or multi-valve repairs/replacements; and
* At University Hospitals Cleveland Medical Center.

Exclusion Criteria:

* Patients with known bleeding disorders, including disseminated intravascular coagulation (DIC), prothrombin deficiency, factor V deficiency, factor VII deficiency, factor X deficiency, factor XI deficiency (hemophilia C), Glanzmann disease, hemophilia A, hemophilia B, idiopathic thrombocytopenic purpura (ITP), and Von Willebrand disease (types I, II, and III);
* Patients undergoing emergent or emergent salvage surgery; and
* Patients actively participating in another clinical trial which could affect outcomes.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Units of Packed Red Blood Cells Transfused | Up to 72 Hours Post-Operative
  Units of packed red blood cells transfused will be measured.
Change in Level of Hematocrit | Baseline, Post-Operative Hours 0, 6, 12, 18, 24, 48, and 72
  Level of hematocrit will be measured at baseline and post-operative.
Change in Level of Plasma Free Hemoglobin | Baseline, Post-Operative Hours 0, 6, 12, 18, 24, 48, and 72
  Level of plasma free hemoglobin will be measured at baseline and post-operative.
Change in Volume of Blood | Baseline, Post-Processing (Up to 120 Minutes)
  Volume of blood will be measured at baseline and post-processing.

SECONDARY OUTCOMES:
Change in Number of Fragmented Red Blood Cells | Baseline, Post-Operative Hours 0, 6, 12, 18, 24, 48, and 72
  Number of fragmented red blood cells will be measured at baseline and post-operative.
Change in Level of Lactate Dehydrogenase | Baseline, Post-Operative Hours 0, 6, 12, 18, 24, 48, and 72
  Level of lactate dehydrogenase will be measured at baseline and post-operative.
Change in Level of Haptoglobin | Baseline, Post-Operative Hours 0, 6, 12, 18, 24, 48, and 72
  Level of haptoglobin will be measured at baseline and post-operative.
Change in Level of Bilirubin | Baseline, Post-Operative Hours 0, 6, 12, 18, 24, 48, and 72
  Level of bilirubin will be measured at baseline and post-operative.
Change in Weight of Surgical Sponge | Baseline, Post-Procedure (Up to 5 Minutes)
  Weight of surgical sponges will be measured at baseline and post-procedure.
Time to Wring Sponges | Up to 120 Minutes
  Time in seconds to wring sponges will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pelletier, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Craig Jarrett, MD, MBA, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No